CLINICAL TRIAL: NCT07080632
Title: An Open Label Clinical Trial to Evaluate the Efficacy and Safety of Calculus Bovis Sativus (CBS) for Intracerebral Hemorrhage
Brief Title: Efficacy and Safety of Calculus Bovis Sativus (CBS) for Intracerebral Hemorrhage(CBSinICH)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Jianmin Pharmaceutical Group Co., LTD. (Industry)
Responsible Party: Principal Investigator, Wei Wang, Professor of Neurology, President of Tongji Hospital, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBSinICH
Record Dates: First submitted 2025-07-10; First posted 2025-07-23 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Intracerebral Hemorrhage; Brain Hemorrhage
Keywords: calculus bovis sativus; Neuroprotection; Neuroinflammation
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages; Neuroinflammatory Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBS therapy, CBS dosage: 300mg per day from day 1 to day 7, in ICH cohort (Experimental): Subjects in ICH cohort of this arm will receive general therapy plus CBS.
  Interventions: Drug: Calculus bovis sativus (CBS)
- NCB therapy,NCB dosage: 300mg per day from day 1 to day 7, in ICH cohort (Experimental): Subjects in ICH cohort of this arm will receive general therapy plus NCB.
  Interventions: Drug: Natural Calculus Bovis(NCB)

INTERVENTIONS:
Drug: Calculus bovis sativus (CBS) — Subjects will orally receive 300mg CBS per day from day 1 to day 7
  Arms: CBS therapy, CBS dosage: 300mg per day from day 1 to day 7, in ICH cohort
Drug: Natural Calculus Bovis(NCB) — Subjects will orally receive 300mg NCB per day from day 1 to day 7
  Arms: NCB therapy,NCB dosage: 300mg per day from day 1 to day 7, in ICH cohort

SUMMARY:
The most common cause of death for Chinese patients is intracerebral hemorrhage(ICH), particularly cerebral infarction. It places a heavy burden on people, families, and society as a whole and poses considerable risks of death and disability. The disease is difficult to identify, and is frequently detected only after it progresses to the point of vascular cognitive dysfunction. The primary ischemia necrosis of brain nerve cells and the activation of inflammatory cells are their pathologic processes.

According to historical Chinese medical documents, bezoar possesses properties that can help prevent seizures, treat strokes, enhance cognitive function and mental well-being, and stimulate alertness. Calculus Bovis Sativus (CBS) is the most authentic formulation of bezoar ingredients compared to other bezoar products. It has received approval from the China Food and Drug Administration for the essential treatment of comatose patients. CBS consists of three primary constituents: bilirubin, bile acids, and taurine. Scientific evidence has demonstrated that all of these components possess anti-inflammatory, antioxidant, and neuroprotective properties.

The investigators' objective is to carry out an investigator-initiated clinical study to assess the efficacy of orally administered CBS in treating intracerebral hemorrhag diseases in humans.

ELIGIBILITY:
Inclusion Criteria:

1. The subject and/or their legal guardian(s) must have full legal capacity, fully understand the purpose, significance, methodology, potential risks, possible adverse effects, types of personal data collected, scope of use, processing methods, retention period, and other relevant information regarding this study. Consent must be given voluntarily.This study will strictly comply with the Personal Information Protection Law, Data Security Law, and other applicable laws/regulations, implementing necessary measures to ensure data security and prevent leakage, tampering, or loss.Upon consent, subjects/guardians authorize the research institution to lawfully process relevant health data, including but not limited to storage, analysis, and statistical use.The institution will strictly limit the scope of personal data usage; no additional purposes will be pursued without separate consent.Subjects/guardians retain the right to access, copy, correct, or delete their data, withdraw consent, or request explanations from the institution.All personal data processing will adhere to legal requirements, ensuring legitimacy, justification, and necessity.
2. Male or female, aged 18-80 years (inclusive) at the time of providing informed nsent.
3. All sexually active participants (male and female of reproductive potential) must use effective contraception during the study and for at least 6 months after the last dose of the investigational treatment.Participants must not donate sperm or eggs during the study or for 6 months post-treatment.
4. Confirmed diagnosis meeting the following criteria:

   1. Hypertensive ICH per Diagnostic Criteria for Spontaneous Intracerebral Hemorrhage in Adults , verified by cranial CT.
   2. Traditional Chinese Medicine (TCM) diagnostic criteria (per Stroke Diagnosis and Efficacy Evaluation Standards by the National TCM Administration's Emergency Research Collaboration Group for Encephalopathy):Primary symptoms: Hemiplegia, impaired consciousness, slurred speech/mutism, sensory deficits, facial deviation.Secondary symptoms: Headache, dizziness, pupillary changes, dysphagia, gaze palsy, ataxia.Diagnosis: ≥2 primary symptoms or 1 primary + 2 secondary symptoms, combined with onset context, predisposing factors, prodromal signs, and age. Imaging may substitute for clinical criteria if insufficient.
   3. Hemorrhage volume: 5-10 mL.
   4. Clinical presentation: Impaired consciousness or significant neurological deficits.
   5. Exclusion: No respiratory failure.
5. Neurological examinations must demonstrate stability within 30 days prior to baseline (Visit 1).

Exclusion Criteria:

1. Medical History and Current Health Status

   1. Any clinically significant history of cardiac, endocrine, hematologic, hepatic, immune, infectious, metabolic, renal, pulmonary, neurological, dermatologic, psychiatric, or other major diseases, as determined by the investigator, that would interfere with trial participation.
   2. Presence of any untreated intracranial tumor at baseline (randomization).
   3. Alternative causes of symptoms, including:Cerebral hemorrhage due to hematologic disorders or bleeding diathesis.Subarachnoid hemorrhage secondary to trauma.Vascular abnormalities (e.g., aneurysms, arteriovenous malformations).Traumatic brain injury, CNS infections, septic encephalopathy, metabolic encephalopathy, epileptic disorders, mitochondrial diseases, Klein-Levin syndrome, Creutzfeldt-Jakob disease, rheumatologic disorders, Reyes syndrome, or inborn metabolic errors.
   4. Any major surgery within 4 weeks before baseline, excluding:

      Laparoscopic or minor procedures (defined as those requiring only local anesthesia/conscious sedation, performed outpatient; e.g., toenail surgery, mole excision, wisdom tooth extraction).Exclusion: Thymoma or teratoma resection.
   5. Planned surgery during the study (except minor procedures).
   6. History of severe allergies/anaphylaxis or any hypersensitivity reaction that may be exacerbated by study treatment components.
   7. Current or history of malignancy (including solid tumors and hematologic malignancies), except:Basal cell/squamous cell carcinoma fully excised and cured ≥12 months before screening.Subjects with cancer in remission for >5 years may be included after sponsor approval.
   8. History of gastrointestinal surgery (except appendectomy/cholecystectomy >6 months before screening), irritable bowel syndrome, inflammatory bowel disease (Crohn's, ulcerative colitis), or other clinically significant active GI disorders.
   9. Clinically significant recurrent/active GI symptoms (e.g., nausea, diarrhea, dyspepsia, constipation) within 90 days before screening, requiring:

      New symptomatic treatment (e.g., GERD medication initiation) or dose adjustments within 90 days.
   10. History of diverticulitis or severe GI abnormalities (e.g., symptomatic diverticulosis) that may increase risks (e.g., perforation).
   11. Blood/plasma/platelet donation (≥1 unit) within 90 days before screening.
   12. Active suicidal ideation within 6 months or suicide attempt within 3 years before screening.
   13. Clinically significant laboratory abnormalities per investigator judgment.
   14. Pregnancy, lactation, or plans to conceive during the study or within 3 months post-treatment.

       Women of childbearing potential must have negative serum/urine pregnancy tests at screening and pre-dose.
   15. Physical/mental conditions compromising safety or efficacy assessments.
   16. Screening/baseline systolic BP >150 mmHg or <90 mmHg after 5-minute rest (one repeat allowed; exclusion if persistent).
   17. Within 3 months before screening:Second-/third-degree AV block, sick sinus syndrome, uncontrolled atrial fibrillation, severe/unstable angina, congestive heart failure, myocardial infarction, or major ECG abnormalities (QTc >450 ms [men] or >470 ms [women; Fridericia correction]).
   18. Planned elective procedures/surgery after ICF signing.
   19. Conditions impairing drug absorption (e.g., gastrectomy).
   20. History of heparin allergy or heparin-induced thrombocytopenia.
   21. Clinically relevant abnormalities in medical history, physical exam, ECG, or lab tests.
2. Infection Risk

   1. HIV infection (positive test/history).
   2. Active hepatitis C (HCV Ab+ with detectable HCV RNA).Allowed: HCV Ab+ with undetectable RNA.
   3. Active hepatitis B (HBsAg+ and/or anti-HBc+).Allowed: Prior natural infection (HBsAg-/anti-HBc+/anti-HBs+) or vaccination (HBsAg-/anti-HBc-/anti-HBs+).
   4. Chronic/severe/recurrent infections (e.g., pneumonia, sepsis) within 90 days before baseline.
   5. TB diagnosis/latent TB (positive IGRA or 2 consecutive tests).
   6. Bacterial/fungal/viral infection symptoms (including URI) within 28 days before baseline Re-screening permitted after successful treatment of localized fungal infections (e.g., candidiasis, tinea).
   7. Infection requiring hospitalization/IV antibiotics within 4 weeks before baseline.
   8. Live/attenuated vaccination within 28 days before baseline or planned during the study.
   9. Contraindications to rescue therapies (rituximab, IVIG, high-dose corticosteroids, IV cyclophosphamide).
   10. Prior treatments:Total lymphoid irradiation, cladribine, T-cell/TCR vaccines, stem cell transplant (any time).
3. Laboratory Values

   1. Clinically significant abnormal lab results at screening/baseline (investigator discretion).
   2. Hematologic abnormalities at screening:

      * WBC <3.0 × 10³/µL
      * ANC <2.0 × 10³/µL
      * Lymphocytes <0.5 × 10³/µL
      * Platelets <100 × 10³/µL
      * ALT/AST/GGT ≥3× ULN or bilirubin >2× ULN
      * eGFR ≤60 mL/min/1.73 m²
      * Lymphocytes <LLN
   3. Urinalysis abnormalities at screening:

      * β-2-microglobulin >0.3 μg/mL
      * Albumin/creatinine ratio >22.6 mg/mmol
4. Other

   1. Prior participation in this study.
   2. Blood donation (≥1 unit) within 90 days, plasma within 1 week, or platelets within 6 weeks before screening.
   3. Alcohol/drug abuse within the past year (investigator-determined).
   4. Pregnancy, lactation, or plans to conceive/breastfeed during the study or within 30 days post-treatment.
   5. Current or prior (within 90 days) participation in another clinical trial.
   6. Clinically significant suicidal ideation/behavior within 12 months (per C-SSRS).
   7. Inability/unwillingness to comply with protocol requirements.
   8. Severe hearing/visual impairment, language barriers, claustrophobia, or other conditions preventing neuropsychological assessments/MRI.
   9. Any other reason deemed by the investigator/sponsor to preclude enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The Modified Rankin Scale (mRS) | Up to 12 weeks after treatment initiation
  To assess mRS of subjects within 12 weeks after treatment initiation. The score ranges from 0 to 5. 5 represents the worst.
National Institute of Health stroke scale (NIHSS) | Up to 12 weeks after treatment initiation
  To assess NIHSS of subjects within 12 weeks after treatment initiation. The score ranges from 0 to 42 represents the worst.
Incidence and Severity of Adverse Effects (AEs) and Severe Adverse Effects (SAEs) | Up to 14 weeks after treatment initiation
  To evaluate the AEs and SAEs occurred within 14 weeks after treatment initiation

SECONDARY OUTCOMES:
Qualitative and quantitative assessment of changes in white matter fiber tracts via brain DTI at Week 12 compared to baseline (Visit 1) and the control group | Up to 12 weeks after treatment initiation
The score of Mini-mental State Examination (MMSE) at week 12 compared with baseline (visit 1) and control group. | Up to 12 weeks after treatment initiation
  The score of MMSE ranges from 0 to 30, and 30 represents the best
Montreal cognitive assessment scale (MoCA) at week 12 compared with baseline (visit 1) and control group. | Up to 12 weeks after treatment initiation
  The score of MoCA ranges from 0 to 30, and 30 represents the best.
The score of Hamilton Anxiety Scale at week 12 compared with baseline (visit 1) and control group. | Up to 12 weeks after treatment initiation
  The score of Hamilton Anxiety Scale ranges from 0 to 56, and 56 represents the worst
The score of Hamilton Depression Scale at week 12 compared with baseline (visit 1) and control group | Up to 12 weeks after treatment initiation
  The score of Hamilton Depression Scale ranges from 0 to 81, and 81 represents the worst
The score of 36-item Short-Form (SF-36) at week 12 compared with baseline (visit 1) and control group | Up to 12 weeks after treatment initiation
  The score of SF-36 ranges from 0 to 100, and 100 represents the best
The incidence of Columbia-Suicide Severity Rating Scale (C-SSRS) events at week 14 compared with baseline (visit 1) and control group. | Up to 14 weeks after treatment initiation

OTHER OUTCOMES:
Qualitative and quantitative changes in MRI（QSM、CEST、DKI） findings at week 12 compared to baseline (Visit 1). | Up to 12 weeks after treatment initiation
Comparison of fecal 16S rRNA sequencing gut microbiota profiles between week 12 and baseline (Visit 1) | Up to 12 weeks after treatment initiation
Comparative analysis of hemorrhagic stress response biomarkers (e.g., inflammatory mediators) in fecal metabolomics between Week 12 and baseline (Visit 1) | Up to 12 weeks after treatment initiation
Profiling of lymphocytes subtypes in serum, including absolute counting and ratio of each type of lymphocyte, at week 12 compared with baseline (visit 1) | Up to 12 weeks after treatment initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei 430000, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang F, Deng Y, Wang H, Fu J, Wu G, Duan Z, Zhang X, Cai Y, Zhou H, Yin J, He Y. Gut microbiota-mediated ursodeoxycholic acids regulate the inflammation of microglia through TGR5 signaling after MCAO. Brain Behav Immun. 2024 Jan;115:667-679. doi: 10.1016/j.bbi.2023.11.021. Epub 2023 Nov 19. PMID 37989444
- [Background] Martinez-Vacas A, Di Pierdomenico J, Gallego-Ortega A, Valiente-Soriano FJ, Vidal-Sanz M, Picaud S, Villegas-Perez MP, Garcia-Ayuso D. Systemic taurine treatment affords functional and morphological neuroprotection of photoreceptors and restores retinal pigment epithelium function in RCS rats. Redox Biol. 2022 Nov;57:102506. doi: 10.1016/j.redox.2022.102506. Epub 2022 Oct 14. PMID 36270186
- [Background] Ohsawa Y, Hagiwara H, Nishimatsu SI, Hirakawa A, Kamimura N, Ohtsubo H, Fukai Y, Murakami T, Koga Y, Goto YI, Ohta S, Sunada Y; KN01 Study Group. Taurine supplementation for prevention of stroke-like episodes in MELAS: a multicentre, open-label, 52-week phase III trial. J Neurol Neurosurg Psychiatry. 2019 May;90(5):529-536. doi: 10.1136/jnnp-2018-317964. Epub 2018 Apr 17. PMID 29666206
- [Background] Liu K, Zhu R, Jiang H, Li B, Geng Q, Li Y, Qi J. Taurine inhibits KDM3a production and microglia activation in lipopolysaccharide-treated mice and BV-2 cells. Mol Cell Neurosci. 2022 Sep;122:103759. doi: 10.1016/j.mcn.2022.103759. Epub 2022 Jul 25. PMID 35901929
- [Background] Jangra A, Gola P, Singh J, Gond P, Ghosh S, Rachamalla M, Dey A, Iqbal D, Kamal M, Sachdeva P, Jha SK, Ojha S, Kumar D, Jha NK, Chopra H, Tan SC. Emergence of taurine as a therapeutic agent for neurological disorders. Neural Regen Res. 2024 Jan;19(1):62-68. doi: 10.4103/1673-5374.374139. PMID 37488845
- [Background] Hurley MJ, Bates R, Macnaughtan J, Schapira AHV. Bile acids and neurological disease. Pharmacol Ther. 2022 Dec;240:108311. doi: 10.1016/j.pharmthera.2022.108311. Epub 2022 Nov 16. PMID 36400238
- [Background] Khalaf K, Tornese P, Cocco A, Albanese A. Tauroursodeoxycholic acid: a potential therapeutic tool in neurodegenerative diseases. Transl Neurodegener. 2022 Jun 4;11(1):33. doi: 10.1186/s40035-022-00307-z. PMID 35659112
- [Background] Li CX, Wang XQ, Cheng FF, Yan X, Luo J, Wang QG. Hyodeoxycholic acid protects the neurovascular unit against oxygen-glucose deprivation and reoxygenation-induced injury in vitro. Neural Regen Res. 2019 Nov;14(11):1941-1949. doi: 10.4103/1673-5374.259617. PMID 31290452
- [Background] Bhargava P, Smith MD, Mische L, Harrington E, Fitzgerald KC, Martin K, Kim S, Reyes AA, Gonzalez-Cardona J, Volsko C, Tripathi A, Singh S, Varanasi K, Lord HN, Meyers K, Taylor M, Gharagozloo M, Sotirchos ES, Nourbakhsh B, Dutta R, Mowry EM, Waubant E, Calabresi PA. Bile acid metabolism is altered in multiple sclerosis and supplementation ameliorates neuroinflammation. J Clin Invest. 2020 Jul 1;130(7):3467-3482. doi: 10.1172/JCI129401. PMID 32182223
- [Background] Liu HW, Gong LN, Lai K, Yu XF, Liu ZQ, Li MX, Yin XL, Liang M, Shi HS, Jiang LH, Yang W, Shi HB, Wang LY, Yin SK. Bilirubin gates the TRPM2 channel as a direct agonist to exacerbate ischemic brain damage. Neuron. 2023 May 17;111(10):1609-1625.e6. doi: 10.1016/j.neuron.2023.02.022. Epub 2023 Mar 14. PMID 36921602
- [Background] Matsui M, Nakanishi T, Noguchi T, Ferrone S. Synergistic in vitro and in vivo anti-tumor effect of daunomycin-anti-96-kDa melanoma-associated antigen monoclonal antibody CL 207 conjugate and recombinant IFN-gamma. J Immunol. 1988 Aug 15;141(4):1410-7. PMID 3135332
- [Background] Thakkar M, Edelenbos J, Dore S. Bilirubin and Ischemic Stroke: Rendering the Current Paradigm to Better Understand the Protective Effects of Bilirubin. Mol Neurobiol. 2019 Aug;56(8):5483-5496. doi: 10.1007/s12035-018-1440-y. Epub 2019 Jan 5. PMID 30612336
- [Background] Vitek L, Tiribelli C. Bilirubin: The yellow hormone? J Hepatol. 2021 Dec;75(6):1485-1490. doi: 10.1016/j.jhep.2021.06.010. Epub 2021 Jun 18. PMID 34153399
- [Background] Zhong XM, Ren XC, Lou YL, Chen MJ, Li GZ, Gong XY, Huang Z. Effects of in-vitro cultured calculus bovis on learning and memory impairments of hyperlipemia vascular dementia rats. J Ethnopharmacol. 2016 Nov 4;192:390-397. doi: 10.1016/j.jep.2016.09.014. Epub 2016 Sep 9. PMID 27616028
- [Background] Lu F, Wang L, Chen Y, Zhong X, Huang Z. In vitro cultured calculus bovis attenuates cerebral ischaemia-reperfusion injury by inhibiting neuronal apoptosis and protecting mitochondrial function in rats. J Ethnopharmacol. 2020 Dec 5;263:113168. doi: 10.1016/j.jep.2020.113168. Epub 2020 Jul 27. PMID 32730869
- [Background] Takahashi K, Azuma Y, Shimada K, Saito T, Kawase M, Schaffer SW. Quality and safety issues related to traditional animal medicine: role of taurine. J Biomed Sci. 2010 Aug 24;17 Suppl 1(Suppl 1):S44. doi: 10.1186/1423-0127-17-S1-S44. PMID 20804621
- [Background] Tang Y, Han Z, Zhang H, Che L, Liao G, Peng J, Lin Y, Wang Y. Characterization of Calculus bovis by principal component analysis assisted qHNMR profiling to distinguish nefarious frauds. J Pharm Biomed Anal. 2023 May 10;228:115320. doi: 10.1016/j.jpba.2023.115320. Epub 2023 Mar 1. PMID 36871364
- [Background] Liu Y, Tan P, Liu S, Shi H, Feng X, Ma Q. A new method for identification of natural, artificial and in vitro cultured Calculus bovis using high-performance liquid chromatography-mass spectrometry. Pharmacogn Mag. 2015 Apr-Jun;11(42):304-10. doi: 10.4103/0973-1296.153083. PMID 25829769
- [Background] Li X, Yao Y, Chen M, Ding H, Liang C, Lv L, Zhao H, Zhou G, Luo Z, Li Y, Zhang H. Comprehensive evaluation integrating omics strategy and machine learning algorithms for consistency of calculus bovis from different sources. Talanta. 2022 Jan 15;237:122873. doi: 10.1016/j.talanta.2021.122873. Epub 2021 Sep 30. PMID 34736706
- [Background] Shimada K, Azuma Y, Kawase M, Takahashi T, Schaffer SW, Takahashi K. Taurine as a marker for the identification of natural Calculus Bovis and its substitutes. Adv Exp Med Biol. 2013;776:141-9. doi: 10.1007/978-1-4614-6093-0_15. PMID 23392879
- [Background] Shi Y, Xiong J, Sun D, Liu W, Wei F, Ma S, Lin R. Simultaneous quantification of the major bile acids in artificial Calculus bovis by high-performance liquid chromatography with precolumn derivatization and its application in quality control. J Sep Sci. 2015 Aug;38(16):2753-62. doi: 10.1002/jssc.201500139. Epub 2015 Jun 30. PMID 26016891
- [Background] Yu ZJ, Xu Y, Peng W, Liu YJ, Zhang JM, Li JS, Sun T, Wang P. Calculus bovis: A review of the traditional usages, origin, chemistry, pharmacological activities and toxicology. J Ethnopharmacol. 2020 May 23;254:112649. doi: 10.1016/j.jep.2020.112649. Epub 2020 Feb 14. PMID 32068140
- [Background] Zhou J, Jiang T, Wang J, Wu W, Duan X, Jiang H, Jiao Z, Wang X. Multimodal investigation reveals the neuroprotective mechanism of Angong Niuhuang pill for intracerebral hemorrhage: Converging bioinformatics, network pharmacology, and experimental validation. J Ethnopharmacol. 2024 Jan 30;319(Pt 1):117045. doi: 10.1016/j.jep.2023.117045. Epub 2023 Aug 24. PMID 37633621